CLINICAL TRIAL: NCT02421965
Title: Comparing Mobile Health (mHealth) and Clinic-Based Self-Management Interventions for Serious Mental Illness: Patient Engagement, Satisfaction, and Outcomes
Brief Title: Comparing Mobile Health (mHealth) and Clinic-Based Self-Management Interventions for Serious Mental Illness
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Dartmouth-Hitchcock Medical Center (Other)
Collaborators: Patient-Centered Outcomes Research Institute (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: STUDY00028548
Record Dates: First submitted 2015-04-16; First posted 2015-04-21 (Estimated); Last update posted 2018-11-20 (Actual); Status verified 2018-11

CONDITIONS: Schizophrenia; Schizoaffective Disorder; Bipolar Disorder; Major Depressive Disorder
Keywords: Schizophrenia; Schizoaffective Disorder; Bipolar Disorder; Major Depressive Disorder; Mobile Application; Smartphone; SMI; Illness Self-Management; EHealth; E-Health; Health Technology; mHealth; m-Health
MeSH Terms: conditions — Schizophrenia; Psychotic Disorders; Bipolar Disorder; Depressive Disorder, Major

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- FOCUS (Smartphone Application) (Experimental): FOCUS is a smartphone application system designed to improve illness self-management and facilitate recovery in individuals with serious mental illness. It delivers both system initiated (i.e. pre-programmed) and patient initiated (i.e. on demand) real-time assessment to individuals in their own environment.
  Interventions: Behavioral: FOCUS (Smartphone Application)
- WRAP (Wellness Recovery Action Planning) (Active Comparator): WRAP is a clinic-based intervention designed to improve illness self-management and facilitate recovery in individuals with serious mental illness. It is conducted in group sessions that are delivered by trained facilitators with lived experience, using lecture, group discussion, and exercises.
  Interventions: Behavioral: WRAP (Wellness Recovery Action Planning)

INTERVENTIONS:
Behavioral: FOCUS (Smartphone Application) — Participants in the FOCUS group will be given a study smartphone device with FOCUS application and trained by the mHealth support specialist on how to use the functions of the smartphone (i.e. using a touchscreen, call, text) and different features of the FOCUS intervention.
  Arms: FOCUS (Smartphone Application)
Behavioral: WRAP (Wellness Recovery Action Planning) — Participants allocated to the WRAP group will be provided all other materials (i.e. WRAP binder, handouts) in their first session and will meet weekly in groups with trained facilitators.
  Arms: WRAP (Wellness Recovery Action Planning)

SUMMARY:
The study is a three year research project whose aims are to evaluate the willingness of individuals with serious mental illness to initiate the two illness self-management interventions- WRAP or FOCUS, to examine and compare participant engagement, satisfaction, and outcomes (symptoms, recovery, quality of life) in the two interventions.

DETAILED DESCRIPTION:
The objective of the study is to compare two illness self-management interventions for SMI: a clinic-based group protocol (Wellness Recovery Action Planning or WRAP) and an mHealth smartphone intervention (FOCUS). The study is structured as a randomized controlled trial, and data will be collected using a comprehensive mixed-methods quantitative /qualitative approach. This study will evaluate patients willingness to enroll in one of the two illness-self management interventions, patient satisfaction, engagement, symptoms, recovery and quality of life.

The specific aims of the study are to: 1) Evaluate and compare the willingness and ability of individuals with SMI to enroll in the two illness self-management interventions; 2) Examine and compare participant engagement and satisfaction with both treatments; and 3) Examine and compare patient outcomes following participation in the interventions.

Participants will be randomized to receive 12-weeks of WRAP or FOCUS. Participants allocated to the WRAP group will be provided all other materials (i.e. WRAP binder, handouts) in their first session and will meet weekly in groups with trained facilitators. Participants in the FOCUS group will be given a study smartphone device with FOCUS application and trained by the mHealth support specialist on how to use the functions of the smartphone (i.e. using a touchscreen, call, text) and different features of the FOCUS intervention.

ELIGIBILITY:
Inclusion Criteria:

* Chart diagnosis of schizophrenia, schizoaffective disorder, bipolar disorder, or major depressive disorder;
* 18 years or older; and
* A rating of "3" or lower on one of the three items which comprise the Domination by Symptoms factor from the Recovery Assessment Scale.

Exclusion Criteria:

* Hearing, vision, or motor impairment that make it impossible to operate a smartphone (determined using demonstration smartphone for screening);
* English reading level below 6th grade (determined using the Wide Range Achievement Test - 4th Edition); and
* Received the FOCUS or WRAP intervention in the past 3 years.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 174 (Actual)
Dates: Start 2015-06; Primary Completion 2017-07 (Actual); Study Completion 2017-12 (Actual)

PRIMARY OUTCOMES:
Patient willingness to enroll / initiate the intervention (WRAP / FOCUS) | 1st day of - attendance of WRAP session OR usage of FOCUS application
  Patient willingness to enroll will be measured by proportion of individuals in each arm who commence the intervention after allocation. It is an important indicator of whether patients find the intervention appealing. Data will be obtained from electronic tracking records / FOCUS software.
Patient Engagement | 3 months
  Patient engagement will be measured by weeks of WRAP sessions attended / weeks FOCUS was used, during the 12-week intervention period. Data for WRAP sessions will be obtained from Thresholds electronic tracking record. Data for FOCUS usage will be captured automatically on FOCUS software.
Patient Satisfaction | 3 months
  Patient satisfaction will be assessed by a 5-item questionnaire on a 7-point scale.
Change in the Severity of Symptoms | Baseline, 3 months (post-treatment), 6 months (follow-up)
  Change in the Severity of Symptoms will measured using Symptom Checklist-9 scale, Beck Depression Inventory-2 (BDI-2) scale and Psychotic Symptom Rating Scale (PSYRATS). Symptom Checklist-9 (SCL-9) is a nine-item questionnaire to assess psychiatric functioning. BDI-2 is a widely used 21-item self-report scale to measure depressive symptom severity. PSYRATS is a fine-grained measure of psychotic symptoms that consists of 17 self-report items that evaluate dimensional symptom severity.
Recovery | Baseline, 3 months (post-treatment), 6 months (follow-up)
  Recovery of patient will be measured using the Recovery Assessment Scale (RAS). RAS has 24 items that assess 5 factors related to recovery including Hope, Goal Directedness, and Domination by Symptoms.
Change in the Quality of Life | Baseline, 3 months (post-treatment), 6 months (follow-up)
  Quality of Life will be assessed using a 6-item Quality of Life scale of general wellbeing, interpersonal relations, participation in activities, and role functioning. Patients respond on a 7-point scale.

CONTACTS AND LOCATIONS:
Overall Officials: Dror Ben-Zeev, PhD, Principal Investigator — Dartmouth Psychiatric Research Center
Locations (1):
- Thresholds Psychiatric Rehabilitation Centers, Chicago, Illinois, United States

REFERENCES:
- [Derived] Ben-Zeev D, Buck B, Chu PV, Razzano L, Pashka N, Hallgren KA. Transdiagnostic Mobile Health: Smartphone Intervention Reduces Depressive Symptoms in People With Mood and Psychotic Disorders. JMIR Ment Health. 2019 Apr 12;6(4):e13202. doi: 10.2196/13202. PMID 30977736
- [Derived] Ben-Zeev D, Brian RM, Jonathan G, Razzano L, Pashka N, Carpenter-Song E, Drake RE, Scherer EA. Mobile Health (mHealth) Versus Clinic-Based Group Intervention for People With Serious Mental Illness: A Randomized Controlled Trial. Psychiatr Serv. 2018 Sep 1;69(9):978-985. doi: 10.1176/appi.ps.201800063. Epub 2018 May 25. PMID 29793397